CLINICAL TRIAL: NCT02193399
Title: Effectiveness of Physiotherapy in the Prevention of Physical Sequelae in Patients Treated With Hematopoietic Stem Cell Transplantation. A Pilot Study.
Brief Title: Physiotherapy in Hematopoietic Stem Cell Transplantation
Acronym: TRAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, RUBÉN CUESTA-BARRIUSO, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRASFIS; TRAS (Other: Universidad Católica San Antonio)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-06

CONDITIONS: Hematologic Malignancy; Stem Cell Transplantation
Keywords: Stem cell transplantation; Fatigue; Physiotherapy; Quality of Life; Cancer; Psychosocial aspects
MeSH Terms: conditions — Hematologic Neoplasms; Fatigue; Neoplasms | interventions — Physical Therapy Modalities; Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy exercises (Experimental): Strength exercises for the muscles proximal upper limbs and lower limbs and proprioception exercises
  Interventions: Other: Physiotherapy in patients with stem cell transplantation
- Control group (No Intervention): Patients undergoing allogeneic transplantation without treatment of physiotherapy

INTERVENTIONS:
Other: Physiotherapy in patients with stem cell transplantation — The exercises are repeated in both upper limbs and both lower limbs. All exercises are performed with specific respiratory exercises simultaneously the movement that takes place each year form.
  The exercises are carried out by the physiotherapist applying in a passive way (ascending or descending) progressive strength and degree of difficulty and variables depending on the clinical condition of the patient.
  Arms: Physiotherapy exercises

SUMMARY:
Research project with patients undergoing allogeneic hematopoietic transplantation in the hematology and hemotherapy Clinical Hospital Universitario Virgen de la Arrixaca. The main objective is to assess the differences in skeletal muscle and functional variables in the experimental group underwent a physiotherapy treatment that takes place during the pre-and post-transplant period, compared to a control group.

DETAILED DESCRIPTION:
The main characteristics of the study are:

* Randomized, prospective and longitudinal in patients receiving allogeneic hematopoietic stem cell transplantation clinical trial.
* A descriptive study of skeletal muscle characteristics of patients undergoing allogeneic hematopoietic transplantation for hematologic malignancies before and after carrying out a treatment with stem cells.
* Clinical study of the variables of strength, mobility, proprioception and upper and lower pain in patients with hematologic malignancy member before and after cancer treatment.
* Clinical study of the effectiveness of physiotherapy treatment in clinical characteristics (strength, mobility, proprioception and pain) in patients undergoing allogeneic stem cell transplantation.
* Clinical study of psychosocial variables that are affected by hematological treatment, and the influence on them of a physiotherapy treatment.

The data obtained in this project to identify and treat those functional deficits that appear as a result of cancer treatment and influencing patients, regarding the evolution of the disease and its treatment. They will use different psychosocial questionnaires and functional tests based on scientific evidence and the reliability of these, as well as its specific design for patients with hematologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years.
* Patients with a diagnosis of hematologic malignancy that will be subjected to hematopoietic transplantation.
* Patients offer sufficient guarantee adherence to protocol.
* Patients who have previously signed informed consent.

Exclusion Criteria:

* Patients with inability to walk, before treatment.
* Patients whose medical judgment contraindicated inclusion in a physiotherapy intervention.
* Patients with psychotic traits, brain damage or senility prevention of the correct understanding of physical therapy.
* Patients with inability to sign informed consent or understanding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Changes in joint range of motion | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days)
  Will be evaluated with a universal goniometer following validated protocols of measurement
Changes in muscle strength of quadriceps, the gastrocnemius and biceps | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  It is measured with the scale of Daniels and a dynamometer.
Changes in proprioception | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  It is measured with a balance platform and supports uni and bipodal
Changes in pain perception | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  It will be evaluated with the visual analogue scale and algometer
Changes in the perception of fatigue | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Using the Spanish version of the Brief Fatigue Inventory
Changes in body mass | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  By using the measurement tool TANITA calculate bone, muscle and fat mass, as well as the amount of fluid of patients at each evaluation.
Changes in the perception of quality of life | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Using the self-questionnaire SF-36 health
Changes in the profile of disease consequences | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Using the questionnaire Sickness Impact Profile (SIP)
Changes in coping with the disease | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Using the scale questionnaire Mental Adjustment to Cancer
Change in perception of anxiety | Screening visit (one month before hospital admission); at the time of admission (±3 days); ±2 days before transplantation; after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Using the STAI questionnaire
Hematopoietic recovery | After hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Measuring the rate of graft failure and the transfusion dependence

SECONDARY OUTCOMES:
Response to the transplantation | After hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  By analyzing the rate and type of response
Infectious complications | After hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  By measuring the rate, type and severity of infections
Noninfectious complications | After hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Measuring the rate of EVOH (number and percentage)
Immunological recovery | after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  By measuring the number and percentage of B lymphocytes, T lymphocytes and NK lymphocytes.
Hospitalisations of the patient after transplantation | after hospital discharge (± 3 days); and at 3 and 6 months after transplantation (± 3 days).
  Measuring the number of hospitalizations, the number of days in hospital and the cause of same
Socio-demographic variables | Screening visit (one month before hospital admission)
  Gender (male, female), academic education (university education, basic education, vocational training), marital status (single, married, divorced, widowed), employment status (self-employed, employed as an employee, unemployed) and distance to hospital (km)
Clinical variables | Screening visit (one month before hospital admission)
  Medical diagnosis, age (years), height (cm), weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: JORGE MONTSERRAT COLL, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia, Spain